CLINICAL TRIAL: NCT05287555
Title: Randomisiert-kontrollierte Klinische Studie an häuslich Beatmeten COPD-Patienten Zur Überprüfung Der Wirksamkeit Einer Telemetrisch unterstützten Fernbetreuung Durch Das Beatmungszentrum im Vergleich Zur stationären, halbjährlichen Beatmungskontrolle gemäß Leitlinie [Randomized-controlled Clinical Trial in Home Ventilated COPD Patients to Test the Efficacy of Telemetry-assisted Care Compared to Biannual Inpatient Ventilation Control Visits According to the Guideline]
Brief Title: Efficacy of Telemetry-assisted Care in Home Home Vented COPD
Acronym: TeleInterVENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georg Nilius, Prof DR med (Industry)
Collaborators: Heinen und Löwenstein GmbH & Co. KG (Industry)
Responsible Party: Sponsor-Investigator, Georg Nilius, Prof DR med, Research and Clinic Director, Institut für Pneumologie Hagen Ambrock eV
Organization: Institut für Pneumologie Hagen Ambrock eV (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TIV2022
Record Dates: First submitted 2022-02-24; First posted 2022-03-18 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; NIV; Telemonitoring
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Prospective, double-arm, controlled-randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Home non-invasive mask ventilation with prisma VENT device. Modem for the daily transmission of specific therapy parameters.
  Standard care according to clinical standard (technical support by the provider and three hospital follow-up appointments after 2, 6 and after 12 months) with assessment of health status and NIV therapy settings.
  Study specific: During visits, recording of HRQOL by SGRQ and S3NIV questionnaires, hospitalizaion and physician visits.
  Therapy data from NIV device.
  Interventions: Other: Standard Care
- Telemonitoring (Experimental): Home non-invasive mask ventilation with prisma VENT device. Modem for the daily transmission of specific therapy parameters. An electronic feedback system provides patients with feedback and recommendations on their therapy based on the data submitted.
  The study center regularly reviews and reacts to all therapy data and other information according to the remote care scheme of intervention.
  Telemonitoring care patients also receive an SpO2 sensor for monitoring of oxygen saturation.
  Ambulantory implementation of three blood gas analyses to check the health status after 2, 6 and 12 months. There are no regular routine inpatient stays.
  Study specific: During visits, recording of HRQOL by SGRQ and S3NIV questionnaires, hospitalizaion and physician visits.
  Interventions: Other: Telemonitoring Care

INTERVENTIONS:
Other: Telemonitoring Care — NIV, Supplies as needed, especially masks, tubes, humidifiers, SpO2 sensor and modems.
  Arms: Telemonitoring
Other: Standard Care — NIV, Supplies as needed, especially masks, tubes, humidifiers, and modems
  Arms: Control

SUMMARY:
This study in patients suffering of Chronic Obstructive Pulmonary disease (COPD) aims to investigate whether telemonitoring of their non invasive ventilation (NIV) device together with targeted, tailored intervention in case of increasing symptoms or ventilation abnormalities improves the therapy adherence and effectiveness and can reduce the need for hospitalizations.

DETAILED DESCRIPTION:
54 NIV naive COPD patients will be randomized to either telemonitoring care with a data-based intervention scheme or standard care according to the guideline of the German Society of Pneumology.

Primary objective:

Adherence to ventilation in the intervention group versus control group.

Secondary objective:

Comparisons between the control and intervention groups, over time and against each other, in terms of:

* Health-related quality of life assessed by SGRQ
* Symptomatology based on blood gas analyses, CAT score, mMRC score and S3-NIV score
* Therapy quality according to therapy parameters from device data
* Number of hospitalizations and physician visits
* Evaluation of the impact of feedback and interventions on therapy adherence, symptomatology and therapy data.

ELIGIBILITY:
Inclusion Criteria:

* NIV-naive / Continuation after 3 Months Interruption
* Indication for initiation of NIV according to S2k guideline of the German Society of Pneumology
* Presence of the signed informed consent

Exclusion Criteria:

* Absence of signed written informed consent for data protection and study participation.
* contraindication to PAP therapy
* Participation in another study that influences the setting of NIV therapy through specifications regarding device settings or titration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-11-24 (Actual)

PRIMARY OUTCOMES:
Adherence [hours/day] | 12 Months
  Usage of Ventilator in hours per day

SECONDARY OUTCOMES:
QOL [unit] | Survey at 3 dates: 2, 6 und 12 Months
  Health related Quality of Life by SGRQ-Score [higher units represent worse outcome]

OTHER OUTCOMES:
Hospitalizations [Nr] | 12 Months
  Number of hospitalizations/physician visits
CAT [score] | Survey at 3 dates: 2, 6 und 12 Months
  COPD Assessment Test, Score 0 to 40, higher units represent worse outcome
mMRC [score] | Survey at 3 dates: 2, 6 und 12 Months
  Modified Medical Research Council, Score 0 to 4, higher units represent worse outcome
S3-NIV [score] | Survey at 3 dates: 2, 6 und 12 Months
  S3-NIV questionnaire for the assessment of home NIV, Score 0 to10, lower units represent worse outcome
PCO2 [mmHg] | Survey at 3 dates: 2, 6 und 12 Months
  Carbon dioxide partial pressure from Blood Gas Analysis

CONTACTS AND LOCATIONS:
Overall Officials: Gearg Nilius, MD, Principal Investigator — KEM | Evang. Kliniken Essen-Mitte gGmbH
Locations (1):
- Evang. Kliniken Essen-Mitte gGmbH, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Time Frame: Starting 6 months and ending 24 months following article publication,
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review commitee identified for this purpose. Proposals may be submitted upt to 24 months following article publication.
URL: https://kem-med.com/kompetenz-in-kliniken/fachkliniken/lungenheilkunde/forschung/